CLINICAL TRIAL: NCT01270373
Title: Randomized Phase II Trial of the Sequences of Anthracyline and Taxane in Locally Advanced Breast Cancer
Brief Title: NeoSAMBA: Neoadjuvant: Does the Sequence of Anthracycline and Taxane Matters: Before or After?
Acronym: NeoSAMBA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, José Bines, MD, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neo2010
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: neoadjuvant therapy; drug therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FAC x 3 followed by Docetaxel x 3 (Active Comparator)
  Interventions: Drug: FAC x 3 followed by Docetaxel x 3
- Docetaxel x 3 followed by FAC x 3 (Experimental)
  Interventions: Drug: Docetaxel x 3 followed by FAC x 3

INTERVENTIONS:
Drug: FAC x 3 followed by Docetaxel x 3 — 5-Fluorouracil (500 mg/m2), Doxorubicin (50 mg/m2) and Cyclophosphamide (500 mg/m2) IV every 21 days, for 3 cycles; followed by Docetaxel 100 mg/m2 every 21 days, for 3 cycles
  Arms: FAC x 3 followed by Docetaxel x 3
Drug: Docetaxel x 3 followed by FAC x 3 — Docetaxel 100 mg/m2 IV every 21 days, for 3 cycles; followed by 5-Fluorouracil (500 mg/m2), Doxorubicin (50 mg/m2) and Cyclophosphamide (500 mg/m2) IV every 21 days, for 3 cycles
  Arms: Docetaxel x 3 followed by FAC x 3

SUMMARY:
The purpose of this study is to evaluate the usual and the reverse sequence of an anthracycline followed by a taxane in locally advanced breast cancer.

DETAILED DESCRIPTION:
Anthracylines and taxanes are the most active chemotherapy agents in the treatment of breast cancer. The usual sequence of an anthracycline followed by a taxane is due to the timing of their discovery and introduction in the treatment armamentarium. More recent evidence suggests that there is pre clinical as well as clinical rational for the reverse sequence.

The neoadjuvant approach allows quick evaluation of these different treatment strategies. At the same time, the study will collect tissue biopsies and blood at different time points in order to evaluate predictive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IIB to IIIB HER-2 negative breast cancer
2. ECOG performance status ≤ 2
3. Neuropathy grade <1 by the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v 3.0)
4. Adequate hematologic function with:

   * Absolute neutrophil count (ANC) >1500/μL
   * Platelets ≥100,000/μL
   * Hemoglobin ≥ 9 g/dL
5. Adequate hepatic and renal function with:

   * Serum bilirubin ≤ 1.5 x the institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x institutional ULN
   * Alkaline phosphatase ≤2.5 x institutional ULN
   * Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥ 50 mL/min
6. Adequate cardiac function

   * Left ventricular ejection fraction (LVEF) within institutional normal range
7. Knowledge of the investigational nature of the study and ability to provide consent for study participation

Exclusion criteria

1. Pregnancy
2. Bilateral, synchronous breast cancer
3. Previous diagnosis of breast or other cancer
4. Any other disease(s), psychiatric condition, metabolic dysfunction, that contraindicates the use of study drugs or that would make the patient inappropriate for this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2010-08; Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 6 months

SECONDARY OUTCOMES:
Cardiac toxicity | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose Bines, MD, Study Chair — INCA Brazil
Locations (1):
- Hospital do Cancer III, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Bines J, Small IA, Sarmento R, Kestelman F, Silva S, Rodrigues FR, Faroni L, Goncalves A, Ebecken E, Maroun P, Millen E, Bonamino M. Does the Sequence of Anthracycline and Taxane Matter? The NeoSAMBA Trial. Oncologist. 2020 Sep;25(9):758-764. doi: 10.1634/theoncologist.2019-0805. Epub 2020 Jun 23. PMID 32476183